CLINICAL TRIAL: NCT02099942
Title: Transluminal Aortic Balloon Valvuloplasty Registry (TAB-R)
Brief Title: Post-Market Surveillance Registry to Monitor Performance and Safety of V8 Device
Acronym: TAB-R
Status: Completed | Type: Observational
Sponsor: InterValve, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1058-001
Record Dates: First submitted 2014-03-18; First posted 2014-03-31 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Balloon Aortic Valvuloplasty; Valvuloplasty; Transcatheter Aortic Valve Replacement; Surgical Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Catheters

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: V8 Balloon Aortic Valvuloplasty (BAV) Catheter — The V8 device can be used for BAV as follows:
  * as stand-alone intervention
  * as a bridge to transcatheter aortic valve replacement (TAVR)
  * as a bridge to surgical aortic valve replacement (SAVR)
  * as an intraprocedural predilatation prior to TAVR

SUMMARY:
This registry is designed to monitor the real world clinical performance and safety of the V8 device used to perform balloon aortic valvuloplasty (BAV). Additional analyses or calculations may be obtained from the imaging or evaluations already performed per the sites' standard of care

DETAILED DESCRIPTION:
The study is an open-label observational study involving a minimum of 10 centers. A minimum of 100 patients, including a minimum of 30 stand-alone balloon aortic valvuloplasty (BAV) treatment patients, will be enrolled. Enrollment will continue until all 3 of these conditions are met.

BAV-only patients will be followed through a 6-month post-treatment telephone follow up. Patients treated with the V8 device for BAV as a bridge to transcatheter aortic valve replacement (TAVR) or surgical aortic valve replacement (SAVR) or as an intraprocedural predilatation prior to TAVR, will exit the study at the time of the TAVR or SAVR implant or at 6 months post-BAV treatment, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic severe aortic stenosis (AS) patients who are not suitable candidates for aortic valve replacement surgery at the time of BAV procedure.
* Subject meets the Indication For Use.
* Probable survival to hospital discharge.
* Subject is competent, willing to comply with evaluations, understands risks, benefits and alternatives and has signed the Informed Consent Form. Alternatively, the legal guardian of the patient is able to give consent to participate.

Exclusion Criteria:

* Patient has undergone previous AVR
* Greater or equal to 3+ aortic insufficiency by echocardiogram obtained prior to planned BAV or intra-procedural predilation TAVR procedure
* Non-valvular AS
* Known congenital AV abnormality (e.g., bicuspid AV)
* Cardiogenic shock, as defined by a consistent systolic blood pressure <80 mmHg off vasopressors or <90 mmHg on vasopressors.
* Bacterial endocarditis ≤ 12 months prior to planned BAV procedure
* Unable to take aspirin (acetyl salicylic acid, ASA) or thienopyridine
* Any illness or condition which, in the Investigator's judgment, will compromise patient safety, or interfere with the interpretation of the treatment results
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic - Patients at each enrolling clinic who are to be treated with the InterValve V8 device for balloon aortic valvuloplasty (BAV) are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Efficacy Endpoint: V8 Device Performance | Intra-procedure
  Successful balloon fixation: proximal and distal balloon segments are securely fixed on either side of the aortic valve annulus following inflation.
Safety Endpoint: Serious Adverse Events (SAE) | Intra-procedure until discharge or 72 hours post-procedure, whichever comes first. (Typical discharge is expected to be within 72 hours.)
  The composite of SAEs as defined by the Valve Academic Research Consortium (VARC).

SECONDARY OUTCOMES:
Efficacy Endpoint: Intra-Procedure Hemodynamic Changes | Intra-procedure
  Absolute and percent change in mean aortic valve (AV) gradient and aortic valve area (AVA).
Efficacy Endpoint: Post-Procedure Hemodynamic Changes | Within 72 hours of procedure or discharge, whichever is first. (Typical discharge is expected to be within 72 hours.)
  Absolute and percent change in mean aortic valve (AV) gradient and aortic valve area (AVA).
Safety Endpoint: Aortic Valve (AV) Block at Discharge | At discharge, which is expected to be within 72 hours procedure.
Safety Endpoint: Aortic Valve (AV) Block at 6-Month Follow-up | 6-Month Follow-up

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Good Samaritin Hospital, Los Angeles, California
  - University of Southern Califormia, Los Angeles, California
  - Abbott Northwestern Hospital (with Minneapolis Heart Institute Foundation), Minneapolis, Minnesota
  - Centennial Heart, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Henrico's Doctors' Hospital, Richmond, Virginia
  - University of Washington, Seattle, Washington